CLINICAL TRIAL: NCT01705054
Title: Angina Prevalence and Provider Evaluation of Angina Relief
Acronym: APPEAR
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IN-US-259-0157
Record Dates: First submitted 2012-09-25; First posted 2012-10-12 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Stable Coronary Artery Disease CAD
Keywords: Angina; Stable ischemic heart disease; Quality of Life; Seattle Angina Questionnaire (SAQ)
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatient Coronary Artery Disease Patient: CAD patients being seen in a participating cardiology office for a scheduled clinic visit who agree to take the survey.

SUMMARY:
The purpose of this study is describe the frequency of chest pain and how chest pain impacts patients' quality of life in the outpatients with chronic coronary artery disease in contemporary cardiology practice settings.

DETAILED DESCRIPTION:
The primary goals in the management of stable coronary artery disease (CAD) are to reduce risk factors for heart attack and to control the symptoms of angina (chest pain). Ideally angina is well controlled with medications alone, but invasive procedures are a valuable option for patients with persistent angina. The amount of angina among patients with stable CAD in the outpatient setting, however, is unknown. An Australian study reported that almost 1 in 3 patients with stable angina being treated by primary care doctors had angina at least once a week, which was associated with worse quality of life. We propose to examine the burden of angina in outpatients with stable CAD who are being medically managed by cardiologists in the United States through administration of a one-time survey. The information from this study could ultimately help improve management of stable CAD and angina and illuminate potential underuse of revascularization. While cardiologists are generally expected to provide better angina control than primary care doctors, establishing the prevalence of angina among the best providers will help with a framework for interpreting symptom control among other practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease patients being seen in a participating cardiology office for a scheduled clinic visit who agree to take the survey.

Exclusion Criteria:

* Too ill to take survey
* Previously completed this survey
* Refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient cardilogy practice.
Sampling Method: Non-Probability Sample
Enrollment: 1246 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07-22 (Actual)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire | One time cardiology office visit.
  Percentage of patients with frequent angina (>1 episode/week) as measured by the Seattle Angina Questionnaire (SAQ).

SECONDARY OUTCOMES:
Quality of Life | One time cardiology office visit.
  Evaluate the impact of frequent angina on Quality of Life (as measured by the SAQ)
Physician Perspective | One time cardiology office visit.
  Identifying differences between patients' and cardiologists' assessment of angina control
Cardiology practices angina control. | One time cardiology office visit.
  Evaluate the differences in angina control between cardiology practices.

CONTACTS AND LOCATIONS:
Overall Officials: John A Spertus, MD, MPH, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri; Faraz Kureshi, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltrame JF, Weekes AJ, Morgan C, Tavella R, Spertus JA. The prevalence of weekly angina among patients with chronic stable angina in primary care practices: The Coronary Artery Disease in General Practice (CADENCE) Study. Arch Intern Med. 2009 Sep 14;169(16):1491-9. doi: 10.1001/archinternmed.2009.295. PMID 19752407